CLINICAL TRIAL: NCT02874534
Title: Development of a Novel Transdiagnostic Intervention for Anhedonia - R61 Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-2268a; R61MH110027-01A1 (NIH)
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-02

CONDITIONS: Anhedonia
MeSH Terms: conditions — Anhedonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Activation (Experimental): Treatment will consist of 15 weekly 45-minute sessions. Session 1 provides orientation and psychoeducation on anhedonia, and activity monitoring is introduced. Sessions 2-3 include structured values assessments of 10 life areas to enhance motivation for sustained behavior change and to clarify goals. Following goals clarification, an activity hierarchy is developed, establishing a set of idiographic behavioral targets across life areas prioritized by ease of implementation to scaffold task engagement during the course of treatment.
  Interventions: Behavioral: Behavioral Activation
- Mindfulness Treatment (Active Comparator): BATA will be compared to mindfulness based cognitive therapy (MBCT), chosen because its mechanisms of action are hypothesized to impact different brain mechanisms than BATA. Mindfulness is nonjudgmentally bringing awareness and acceptance to one's present-moment experience. MBCT will be administered in an individual format. The MBCT protocol will be modeled on the session outlines presented in Wahbeh et al., 2014. Treatment will be compromised of 15 weekly 45-minute sessions.
  Interventions: Behavioral: Mindfulness Treatment

INTERVENTIONS:
Behavioral: Behavioral Activation — Treatment will consist of 15 weekly 45-minute sessions.
  Arms: Behavioral Activation
Behavioral: Mindfulness Treatment — Treatment will consist of 15 weekly 45-minute sessions.
  Arms: Mindfulness Treatment

SUMMARY:
The overall goal of this project is to develop a novel transdiagnostic treatment for anhedonia, called Behavioral Activation Treatment for Anhedonia (BATA), using ultra-high field functional neuroimaging. There is a critical need for a validated treatment that specifically targets anhedonia, and this project will evaluate the effects of this new treatment on anhedonia and will establish how this treatment impacts brain systems that mediate reward processing, clinical symptoms of anhedonia, functional outcomes, and behavioral indices of reward processing. This work will also identify brain targets by which future novel anhedonia treatment may be evaluated.

DETAILED DESCRIPTION:
Deficits in motivation and pleasure, together referred to as anhedonia, are implicated in a number of psychiatric illnesses, including mood and anxiety disorders, substance-use disorders, schizophrenia, and attention-deficit/hyperactivity disorder. As a result, constructs related to anhedonia are central to the NIMH Research Domain Criteria (RDoC) project. Anhedonia is often one of the most difficult psychiatric symptoms to treat and thus represents a critical endophenotype and vulnerability factor for a range of psychiatric disorders. Given the centrality of anhedonia to a large number of psychiatric disorders, improved interventions to treat motivation and pleasure are critical for these disorders. The overall goal of this R61/R33 project is to develop a novel transdiagnostic treatment for anhedonia, called Behavioral Activation Treatment for Anhedonia (BATA). This new intervention is designed to treat anhedonia by emphasizing supported engagement with personally relevant goals and reducing avoidance behaviors. Consistent with the objectives and milestones outlined in RFA-MH-16-406 ("Exploratory Clinical Trials of Novel Interventions for Mental Disorders"), in the R61 phase of this trial that lasted from June 22, 2017-July 31, 2019, the investigators propose to use an experimental therapeutics approach to first evaluate mesocorticolimbic target engagement by this treatment in a transdiagnostic sample characterized by clinically impairing anhedonia (Aim 1). Specifically, the investigators will examine the effects of this treatment, relative to an active comparison treatment, on caudate nucleus activation during reward anticipation and rostral anterior cingulate cortex activation during reward outcomes using ultra-high field (7T) functional magnetic resonance imaging. In this phase of the project, the investigators will also use fMRI to determine the optimal dose of the intervention (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

1. 18-50 years old and treatment seeking;
2. SHAPS scores ≥ 20, corresponding to clinically significant anhedonia;
3. Clinician's Global Impression Scale-Severity score (CGI-S) > 3 to assure a clinically impaired sample;
4. Seeking treatment for anhedonia (i.e., referred from an outpatient clinic or responded to an advertisement for anhedonia treatment; endorses desire for treatment during screening).

Exclusion Criteria:

1. Those for whom medication management is the primary gold-standard treatment, including those with bipolar disorder/mania, schizophrenia spectrum, and other psychotic disorders;
2. Prior treatment with behavioral activation therapy for depression or mindfulness-based treatments (those with exposure to other forms of psychotherapy, e.g., supportive therapy, will be eligible);
3. Those who may have difficulty understanding the cognitive components of BATA, including those with intellectual disability, neurocognitive disorders, and dissociative disorders;
4. Feeding and eating disorders which may have confounding effects on the fMRI signal;
5. Substance Use Disorders given confounding effects of substances of abuse on the fMRI signal;
6. Suicidal intent and plan;
7. Psychotropic medication use in the past 4 weeks (8 weeks for fluoxetine) and/or current psychotherapy. Participants must be medication-free at study entry; study personnel will not supervise medication taper for the purpose of the study, but those who taper under the supervision of their regular provider will be eligible;
8. Currently pregnant, as measured by urine pregnancy screen immediately before MRI scans;
9. Positive urinalysis screen for cocaine, marijuana, opiates, methadone, amphetamines, and benzodiazepines (conducted on-site via Biosite Triage Meter Plus) at study entry.
10. No neurological conditions (e.g., history of stroke, seizure, or TBI);
11. Contraindications for fMRI imaging: Metal in the body, dental work that is not fillings or gold, any tattoos, any metal in the body, any metal injury - especially those to the eyes, any other type of implant unless they are 100% plastic.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel S Dichter, PhD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via the NIMH Data Archive (NDA), collection #2595. Investigators may access the deidentified IPD directly from NDA without needing to contact the study team directly.
Time Frame: Time Frame: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication.
Access Criteria: To request access to data, you must be sponsored by an NIH-recognized institution with a Federalwide Assurance and have a research related need to access NDA data. See https://nda.nih.gov/get/access-data.html for more information.
URL: https://nda.nih.gov/edit_collection.html?id=2595

REFERENCES:
- [Derived] Cernasov PM, Walsh EC, Nagy GA, Kinard JL, Kelley L, Phillips RD, Pisoni A, Diehl J, Haworth K, West J, Freeman L, Pfister C, Scott M, Daughters SB, Gaylord S, Dichter GS, Smoski MJ. A parallel-arm, randomized trial of Behavioral Activation Therapy for anhedonia versus mindfulness-based cognitive therapy for adults with anhedonia. Behav Res Ther. 2024 Nov;182:104620. doi: 10.1016/j.brat.2024.104620. Epub 2024 Aug 23. PMID 39213738
- [Derived] Gibson K, Cernasov P, Styner M, Walsh EC, Kinard JL, Kelley L, Bizzell J, Phillips R, Pfister C, Scott M, Freeman L, Pisoni A, Nagy GA, Oliver JA, Smoski MJ, Dichter GS. The effects of psychotherapy for anhedonia on subcortical brain volumes measured with ultra-high field MRI. J Affect Disord. 2024 Sep 15;361:128-138. doi: 10.1016/j.jad.2024.05.140. Epub 2024 May 28. PMID 38815760
- [Derived] Cernasov PM, Kinard JL, Walsh E, Kelley L, Phillips R, Pisoni A, Arnold M, Lowery SC, Ammirato M, Nagy GA, Oliver JA, Haworth K, Daughters SB, Dichter GS, Smoski M. Parsing within & between-person dynamics of therapy homework completion and clinical symptoms in two cognitive behavioral treatments for adults with anhedonia. Behav Res Ther. 2023 Jul;166:104322. doi: 10.1016/j.brat.2023.104322. Epub 2023 Apr 26. PMID 37148652
- [Derived] Phillips R, Walsh E, Jensen T, Nagy G, Kinard J, Cernasov P, Smoski M, Dichter G. Longitudinal associations between perceived stress and anhedonia during psychotherapy. J Affect Disord. 2023 Jun 1;330:206-213. doi: 10.1016/j.jad.2023.03.011. Epub 2023 Mar 11. PMID 36907457

RESULTS

PARTICIPANT FLOW:
Groups:
- Mindfulness Treatment: Behavioral Activation Treatment for Anhedonia (BATA) will be compared to mindfulness based cognitive therapy (MBCT), chosen because its mechanisms of action are hypothesized to impact different brain mechanisms than BATA. Mindfulness is nonjudgmentally bringing awareness and acceptance to one's present-moment experience. MBCT will be administered in an individual format. The MBCT protocol will be modeled on the session outlines presented in Wahbeh et al., 2014. Treatment will be compromised of 15 weekly 45-minute sessions.
  Mindfulness Treatment: Treatment will consist of 15 weekly 45-minute sessions.
Period: Overall Study
Arm/Group | Behavioral Activation | Mindfulness Treatment
Started | 31 | 26
Completed | 23 | 15
Not Completed | 8 | 11
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Lost to Follow-up | 2 | 2
Not completed — Ongoing in study | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Activation | Mindfulness Treatment | Total
Number analyzed (Participants) | 31 | 26 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.61 (8.47) | 33.35 (9.25) | 30.23 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 18 | 16 | 34
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 26 | 57
SHAPS [Mean (Standard Deviation); unit: units on a scale] — The Snaith-Hamilton Pleasure Scale (SHAPS) is a 14-item self-report scale that measures the ability to experience pleasure. The SHAPS scale has a range from 14-56. Higher scores on the SHAPS scale indicate less ability to experience pleasure.
  units on a scale | 37.61 (4.38) | 38.00 (5.25) | 37.79 (4.76)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 15 in Neural Activation
Description: Change due to BATA, relative to MBCT, from baseline in right caudate nucleus activation during the anticipation phase of the Monetary Incentive Delay (MID) task assessed by Functional Magnetic Resonance Imaging (fMRI). The BOLD (Blood Oxygen Level-Dependent signal change is expressed as a z-score that represents the magnitude of change relative to baseline. A score of 0 would correspond to no change, and a score of 1 would represent 1 standard deviation of change. The difference in z-scores between the BATA and the MBCT groups reflects the difference in change in fMRI responses between the two treated groups. Thus even a score of 0 in the BATA group may reflect greater change than observed in the MBCT group if change in the MBCT group is negative.
Time Frame: Baseline, 15 weeks
Population: The fMRI data quality for one participant was inadequate and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Behavioral Activation | Mindfulness Treatment
Number analyzed (Participants) | 22 | 15
Z-score | 0.0075 (0.23) | -0.1059 (0.21)

2. Secondary Outcome: Change From Baseline to Week 15 in Snaith-Hamilton Pleasure Scale Score
Description: The Snaith-Hamilton Pleasure Scale (SHAPS), used to assess hedonic capacity. The sum of the 14 items scores ranges from 0 to 56. A higher score represents more anhedonic symptoms. The below means represent change in units on the Snaith-Hamilton Pleasure Scale.
Time Frame: Baseline, 15 weeks
Population: The fMRI data quality for one participant was inadequate and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Activation | Mindfulness Treatment
Number analyzed (Participants) | 22 | 15
units on a scale | 8.0 (4.87) | 9.3 (7.6)

ADVERSE EVENTS:
Time Frame: From initial assessment through post treatment scan, a total of approximately 3 to 5 months.
Description: Study team members (e.g., study coordinator, study therapists) asked participants at each visit following the initial appointment if any adverse events or changes in health were experienced since the last visit. Adverse Events were assessed by a trained study coordinator, study therapist, or other approved study team member, and discussed at the weekly research staff meetings.
Arm/Group | Behavioral Activation | Mindfulness Treatment
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/26
Other Adverse Events (participants affected / at risk) | 10/31 | 12/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Activation (N=31) | Mindfulness Treatment (N=26)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Burns on right forearm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cold Symptoms (Infections and infestations) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Elevated TSH (Endocrine disorders) | 0 (0) | 1 (1)
Flu (Infections and infestations) | 0 (0) | 1 (1)
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Intermittent eye twitching (Eye disorders) | 1 (1) | 0 (0) — Intermittent eye twitching after mri scan
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Scalp Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sinus Infection (Infections and infestations) | 2 (2) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) — Suicidal Ideation secondary to motor vehicle accident
Telogen Effluvium (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Presyncopal Episode (Cardiac disorders) | 0 (0) | 1 (1)
Broken Collar Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Streptococcal pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Worsening arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — worsening arthritis pain (back & neck) secondary to MRI

LIMITATIONS AND CAVEATS:
These results represent the complete therapeutic target results for this trial's R61 phase that may be combined with the results of the ongoing clinical endpoint R33 phase study whose final results will be reported in NCT04036136.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT02874534/Prot_SAP_000.pdf